CLINICAL TRIAL: NCT05595031
Title: Evaluation of the Clinical Impact of Corticosteroid Duration on SARS-CoV-2 Acute Respiratory Distress Syndrome
Brief Title: Evaluation of the Clinical Impact of Corticosteroid Duration on SARS-CoV-2 (COVID-19 WHO)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Methodist Health System (Other)
Responsible Party: Sponsor
Other Study IDs: 044.PHA.2021.D
Record Dates: First submitted 2022-05-24; First posted 2022-10-26 (Actual); Last update posted 2022-10-26 (Actual); Status verified 2022-10

CONDITIONS: Covid 19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this project is to evaluate the clinical impact of the use of glucocorticoids beyond 10 days for patients with critical COVID-19 at MDMC.

DETAILED DESCRIPTION:
The purpose of this project is to evaluate the clinical impact of the use of glucocorticoids beyond 10 days for patients with critical COVID-19 at MDMC.

Glucocorticoids have become standard of care for critical COVID-19 patients, with a mortality benefit shown in several recent randomized control trials. Critical COVID-19 can lead to ARDS, in which the use of glucocorticoids has uncertain benefit beyond 10 days. Studies have shown increased harm in the use of these agents in persistent ARDS (≥14 days). Additionally, studies supporting the use of steroids in COVID-19 only used steroids for a limited time (up to 10 days). Given that these agents can possibly lead to increased patient morbidity and mortality, prolonged use of glucocorticoids is not without risk. To date, there have been no studies evaluating the clinical impact of glucocorticoid use beyond 10 days for treatment of critical COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years of age
* ICU admission at any time during first hospital admission for COVID-19
* COVID-19 diagnosis
* Dexamethasone, hydrocortisone, or methylprednisolone therapy for SARS-CoV-2 infection

Exclusion Criteria:

* Prior ICU admission before study start date
* Death or hospice before day 11 of hospital admission
* Still admitted at time of data analysis from index admission

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a retrospective chart review study limited to only patients meeting inclusion and exclusion criteria. Determination of the clinical impact of corticosteroid dosing will be aided by a larger cohort of patients. We plan to conduct the retrospective chart review of all patients identified during the study period 08/01/2020 to 01/31/2021 that meet inclusion and exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2021-10-19 (Actual); Primary Completion 2023-10-19 (Estimated); Study Completion 2023-10-19 (Estimated)

PRIMARY OUTCOMES:
All-cause in-hospital mortality at 28 days | 28 days
  All-cause in-hospital mortality at 28 days

SECONDARY OUTCOMES:
Bacteremia | 28 days
  growth of a pathogenic organism in 1 of 4 blood culture sites; blood cultures are considered contaminants if 1 of 4 sets grows a typically non-pathogenic organism or if the clinical team determines the organism a contaminant. To determine if the use of corticosteroids beyond 10 days increases the incidence of secondary infection or impacts duration of MV and length of stay in critical COVID-19.
Mechanical ventilator-free days | 28 days
  number of days alive and breathing without assistance
ICU LOS | 28 days
  number of days alive and admitted to the ICU
Hospital LOS | 28 days
  number of days alive and admitted to MDMC
hospital acquired pneumonia (HAP) | 28 days
  New lung infiltrate after 48 hrs of admission, positive respiratory culture, AND clinical evidence suggestive of new infection. To determine if the use of corticosteroids beyond 10 days increases the incidence of secondary infection or impacts duration of MV and length of stay in critical COVID-19.
ventilator-associated pneumonia (VAP) | 28 days
  VAP arises >48 hrs after intubation. To determine if the use of corticosteroids beyond 10 days increases the incidence of secondary infection or impacts duration of MV and length of stay in critical COVID-19.
C. diff infection (CDI) | 28 days
  Acute onset of diarrhea (> 3 unformed or watery stools occurring in < 24 hours) AND positive test for toxigenic C. difficile or pseudomembranous colitis on endoscopy OR high clinical suspicion. To determine if the use of corticosteroids beyond 10 days increases the incidence of secondary infection or impacts duration of MV and length of stay in critical COVID-19.

CONTACTS AND LOCATIONS:
Overall Officials: Kristen Rahmanzadeh, PharmD, Principal Investigator — The Methodist Hospital Research Institute
Locations (1):
- Methodist Dallas Medical Center, Dallas, Texas, United States